CLINICAL TRIAL: NCT04567251
Title: Survivorship Study of Cancer Patients Who Received Cranial Radiation Therapy: Focus on Health-Related Quality of Life and Cognition
Brief Title: Survivorship Study of Cancer Patients Who Received Cranial Radiation Therapy
Acronym: SPiRiT
Status: Terminated | Type: Observational
Why Stopped: PRMC closed for low accrual
Sponsor: Duke University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00102684
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Brain Metastases, Adult; Primary Brain Tumor; Lung Cancer
Keywords: Pro00102684; Katherine Peters; Lung Cancer; Brain metastases; Brain tumor; Radiation; Solid tumor; Cognition; Pediatric Cancer; Cancer Survivor; Survivorship; Noona; Healthcare Mobile Application
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Noona® mobile healthcare application: All patients will be instructed to report pre-defined, non-life-threatening cognitive symptoms as often as relevant through the Noona® application for 17 weeks.
  Interventions: Other: Noona® application

INTERVENTIONS:
Other: Noona® application — A digital symptom tracking application focused on Health-Related Quality of Life (HRQOL) and cognition in cancer survivors who received brain irradiation

SUMMARY:
This study represents a survivorship protocol that focuses on cognition and health-related quality of life (HRQoL) in cancer patients that have received prior brain irradiation. The primary purpose of this study is to assess the feasibility of using a digital symptom tracking application focused on HRQoL and cognition in cancer survivors who received brain irradiation.

DETAILED DESCRIPTION:
Patients who may participate in the study are cancer survivors who received cranial irradiation for conditions including, but not limited to: primary brain tumors, brain metastases, patients with lung cancer receiving prophylactic brain irradiation, and long-term survivors of pediatric cancers. Patients will use the Noona® Healthcare Mobile PRO Application to identify real time select HRQoL and cognitive symptoms. Patients will be instructed to log symptoms as often as relevant using their own personal devices, as well as be prompted to fill out the Patient-Reported Outcomes Measurement Information System Global Health Screen (PROMIS Global Health-10 and Edmonton Symptom Assessment Scale) during treatment (weeks 9 and 14). Patient engagement with the application will be tracked to determine feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer survivors who received cranial irradiation including, but not limited to, primary brain tumor, brain metastases, lung cancer receiving prophylactic brain irradiation, long-term survivors of pediatric cancers
2. Initial radiation must have been completed more than 6 months prior to enrollment. Acceptable radiation therapies include fractionated partial brain irradiation, whole brain irradiation, or stereotactic radiosurgery (for any modality at least a total cumulative dose of 20 Gy) of at least 20 Gy
3. Age ≥ 18 years at the time of entry into the study
4. Karnofsky performance score (KPS) ≥ 70 or Eastern Cooperative Oncology Group (ECOG) grade ≤ 2
5. No imaging evidence of disease progression within 4 months of enrollment
6. Life expectancy > 6 months per treating neuro-oncology providers
7. Access to a smartphone, tablet, or computer with capability to utilize the mobile symptom-tracking application
8. Subject must be fluent in English

Exclusion Criteria:

1. Active psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer survivors who received cranial irradiation including, but not limited to, primary brain tumor, brain metastases, lung cancer receiving prophylactic brain irradiation, long-term survivors of pediatric cancers
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of using a digital symptom tracking application focused on HRQoL and cognition in cancer survivors who received brain irradiation | Baseline, 15 weeks
  The percentage of patients returning for their Week 15 clinic appointment who initiate PROMIS and ESAS questionnaires via the mobile application at Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Duke Health Clinical Trials — https://www.dukehealth.org/clinical-trials
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/